CLINICAL TRIAL: NCT05813249
Title: Therapeutic Effect of Semaglutide on Nonalcoholic Fatty Liver Disease in Obesity and/or Type 2 Diabetes Mellitus
Brief Title: Semaglutide in Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ayman Magd Eldin Mohammad Sadek, Associate Professor of Internal Medicine, Zagazig University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB#10461/15-2-2023
Record Dates: First submitted 2023-03-19; First posted 2023-04-14 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Semaglutide; Non-alcoholic Fatty Liver Disease; Obesity; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NAFLD1 (Active Comparator): Hepatic steatosis
  Interventions: Drug: Rybelsus Oral Product
- NAFLD2 (Active Comparator): Hepatic steatosis
  Interventions: Drug: Ozempic Injectable Product
- NAFLD3 (Active Comparator): Hepatic steatosis
  Interventions: Drug: Tocopherol and/or Actos

INTERVENTIONS:
Drug: Rybelsus Oral Product — Oral Semaglutide
  Arms: NAFLD1
Drug: Ozempic Injectable Product — Subcutaneous Semaglutide
  Other Names: Wegovy
  Arms: NAFLD2
Drug: Tocopherol and/or Actos — Vitamin E and/or Pioglitazone
  Arms: NAFLD3

SUMMARY:
The goal of this clinical trial is to test the therapeutic effect of Semaglutide in NAFLD and its sequelae in obesity and/or type 2 diabetes mellitus. The main question it aims to answer is:

• Is the use of Semaglutide (oral or subcutaneous form) effective in improving NAFLD and its sequelae in obesity and/or type 2 diabetes mellitus?

Participants will undergo:

* Abdominal ultrasound.
* Fibroscan with controlled attenuation parameter to assess liver stiffness (kPa) and liver steatosis (dB/m).
* Fibrosis-4 score requires values of age, alanine aminotransferase, aspartate aminotransferase, and platelet count.
* NAFLD Fibrosis Score requires values of age, BMI, platelet count, albumin, hyperglycemia, and ALT/AST ratio.

Researchers will compare:

* Group 1 will receive oral Semaglutide for 48 weeks.
* Group 2 will receive injectable Semaglutide for 48 weeks.
* Group 3 will receive Pioglitazone and/or Vitamin E. to see if there is an improvement in liver stiffness and severity of hepatic steatosis after 48 weeks.

DETAILED DESCRIPTION:
Rationale:

NAFLD is one of the major causes of chronic liver disease worldwide with the highest prevalence in Middle East countries. No pharmaceutical agent until now approved to treat hepatic steatosis. There is a potential effect of glucagon-like peptide-1 agonists in the treatment of steatosis and improving the resulting steatohepatitis and fibrosis in obesity and/or type 2 diabetes mellitus.

Research question:

Is the use of Semaglutide (oral or SC form) effective in improving NAFLD and its sequelae in obesity and/or type 2 diabetes mellitus?

Hypothesis:

The investigators hypothesize that Semaglutide (oral or SC form) has a role in NAFLD associated with obesity and/or type 2 diabetes mellitus.

Aim of the study:

To determine the therapeutic effect of Semaglutide in NAFLD and its sequelae in obesity and/or type 2 diabetes mellitus.

Objectives:

* Determine the therapeutic effect of oral and SC Semaglutide in NAFLD and its sequelae in obesity and/or type 2 diabetes mellitus.
* Compare oral and SC forms of Semaglutide.
* Evaluate the impact of the medication on glycemic control and weight loss.

Material and methods:

1. Site of study:

   This study will be conducted in Internal Medicine Department, at Zagazig University Hospitals.
2. Type of study:

   This study is an open-label clinical trial.
3. Subjects allocation:

   * Group 1: patients receive oral Semaglutide for NAFLD complicating obesity and/or type 2 diabetes.
   * Group 2: patients receive SC Semaglutide for NAFLD complicating obesity and/or type 2 diabetes.
   * Group 3: patients receive conventional drug therapy for NAFLD (vitamin E and/or pioglitazone) complicating obesity and/or type 2 diabetes.
   * The patients receive medication at their own expense from a private pharmacy.
4. Steps of performance and techniques:

   * Full medical history taking.
   * Complete physical examination for all patients, calculating body mass index.
   * Local examination of the liver.
   * Calculation of BMI and measurement of waist circumference.
   * Liver function tests.
   * Complete blood count.
   * Kidney function tests.
   * Lipid profiles include total cholesterol, triglyceride, LDL, and HDL.
   * Glucose metabolisms include fasting plasma glucose and HbA1c.
   * Abdominal ultrasound.
   * Fibroscan with CAP to assess liver stiffness (kPa) and liver steatosis (dB/m).
   * FIB4 requires values of age, ALT, AST, and platelet count.
   * NFS requires values of age, BMI, platelet count, albumin, hyperglycemia, and ALT/AST ratio.
   * Group 1 will receive oral Semaglutide with starting dose of 3mg daily then up-titration to 14 mg for 48 weeks. Group 2 will receive injectable Semaglutide starting with 0.25mg SC weekly for 4 weeks and up-titration gradually to reach 2mg SC weekly for 48 weeks. Group 3 will receive Pioglitazone and/or Vitamin E.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with NAFLD by non-invasive methods in the form of abdominal US or MRI, confirmed by a Fibroscan scan with CAP to assess the quantity of hepatic steatosis and severity of fibrosis up to 21 weeks before the start of the study and after treatment.
* Primary obesity with body mass index (BMI) > 30.
* Type 2 diabetes mellitus.

Exclusion Criteria:

* Type 1 diabetes mellitus.
* DM, which is treated with insulin glargine.
* Alcohol consumption.
* Patients had bariatric surgery.
* Hepatitis C virus, hepatitis B virus, HIV.
* Patients with peptic ulcer disease.
* Secondary obesity originated from hypothalamic or endocrinal disorders.
* Other causes of CLD.
* Decompensated liver disease.
* History of pancreatitis (acute or chronic).
* Hepato-biliary disorders.
* ALT and AST values > 5 times of upper normal limits.
* Severe cardiac disease.
* Patients treated with GLP-1 agonist within 90 days before screening.
* Patients with a personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
NAFLD regression | 48 weeks
  improvement of severity of hepatic steatosis evaluated by CAP (dB/m)

SECONDARY OUTCOMES:
Fibrosis regression | 48 weeks
  improvement of liver stiffness evaluated by Fibroscan (kPa) and

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Sadek, MD, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No